CLINICAL TRIAL: NCT05495802
Title: Regional Database for Collecting Clinical-biological and Imaging Data "Secondary Bone Oncology and Bone Localizations of Hematologic Diseases"
Acronym: OOSLOH
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Lille University Hospital Emergence Fund (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019_59; 2021-A00829-32 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-08-03; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Bone Metastases
Keywords: bone localisations of haematological diseases; Cancer; bone metastasis; haematological diseases; quality of life; epidemiological data
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Improving the effectiveness of cancer treatments makes it possible to lengthen patient survival. It is therefore important to ensure that the quality of life is also maintained by reducing pain and handicap.

Some cancers tend to spread to the bone. The bone locations of cancer can weaken the bone and lead to complications such as fractures, pain, or compression of neurological structures.

To avoid such complications, weekly multidisciplinary meetings (MM) bring together specialists (oncologists, rheumatologists, cancer surgeons, radiologists, radiotherapists, etc.) to discuss the files of patients with bone lesions from cancer. They offer specific treatments adapted to each patient to treat or reduce the risk of complications. The OOSLOH study aims to collect clinical, biological, and imaging data from patients for whom a discussion took place in bone dedicated MM. Based on these data, epidemiological studies could be carried out to better understand the clinical factors leading cancer to colonize bone. But also to determine the factors making it possible to prevent or better treat bone complications and improve the quality of life of patients. This study does not require any examinations or additional visits to the patient

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over,
* Patient whose file is presented to the OOSLOH MM and who has not objected to the use of his non-nominative clinical, biological and imaging data
* Social insured patient

Exclusion Criteria:

* Patient who died before presentation to OOSLOH MM,
* Minor patient,
* Patient objecting to the use of their data for research purposes,
* Patient unable to express his right to object to his participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients whose file is presented in MM OOSLOH for a diagnostic, therapeutic or follow-up question of a malignant bone lesion
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2032-11 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of alive patients | through study completion, an average of 10 years

SECONDARY OUTCOMES:
Percentage of patients without bone disease recurrence | within one year after the multidisciplinary meeting
Time to bone disease recurrence | through study completion, an average of 10 years
Number of bone recurrence Number of bone recurrence | At each presentation of the patient file's to the MM,on average every week
Epidemiological datas | At the first presentation of patient's file to the MM, on average every week

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Hélène VIEILLARD, MD, Principal Investigator — University Hospital, Lille